CLINICAL TRIAL: NCT04726540
Title: A Seven-year Follow-up Study of Patient Satisfaction With Three-Implant-Retained Mandibular Overdentures
Status: Completed | Type: Observational
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Hisham ElGabry, Ass. Prof. Prosthodontics, October University for Modern Sciences and Arts
Other Study IDs: 1224
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Patient Satisfaction Using Implant Retained Overdentures
Keywords: patient satisfaction,implant-retained overdenture,complete denture
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I
  Interventions: Other: Patient Satisfaction
- Group II
  Interventions: Other: Patient Satisfaction

INTERVENTIONS:
Other: Patient Satisfaction — Patients were then asked to grade their overdentures/dentures on a visual analog scale and written questionnaire to evaluate their overall satisfaction.

SUMMARY:
Purpose: This study aimed to compare patients' satisfaction with mandibular overdentures retained by three-splinted implants and conventional complete dentures during a seven-year follow-up period. Materials and Methods: Thirty edentulous male patients (mean age: 60 years) were carefully selected and divided into two equal groups. All patients received a new set of complete dentures. (Group I) patients received three implants in the anterior mandible and were connected after three months with bars, clips and loaded. (Group II) patients' received conventional complete dentures. Patients' satisfaction was recorded for both groups at three weeks (baseline) and after 1, 3, 5 and 7 years. Patients were then asked to grade their overdentures/dentures on a visual analog scale and written questionnaire to evaluate their overall satisfaction. Results: satisfaction scores of Group I patients was found to be statistically significantly higher than that of Group II patients (p < .05) at 3, 5 and 7 years follow-up, meanwhile no statistically significant difference was found at baseline or after 12 months. Conclusions: The long-term results suggest that three implants-retained mandibular overdenture with a clip-bar attachment appears to be a successful rehabilitation strategy which is superior to conventional dentures for patients with advanced ridge resorption.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria stipulated that patients must have been wearing dentures on a regular basis, have been edentulous for a minimum of 3-years, and are capable of reading and writing.

Exclusion Criteria:

* insufficient bone volume to install three 13mm. interforaminal implants (Group I), insufficient interarch space. Patients with diabetes, osteoporosis, smokers, psychological problems of removable denture acceptance, gag reflex, absence of a maxillary complete denture and medical or physical considerations that would seriously affect the surgical procedure (Group I) or the follow-up period were also excluded

Ages: 58 Years to 62 Years | Sex: Male
Age Groups: Adult
Study Population: patients must have been wearing dentures on a regular basis, have been edentulous for a minimum of 3-years, and are capable of reading and writing.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01-12 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Seven years
  Patients were then asked to grade their overdentures/dentures on a visual analog scale and written questionnaire to evaluate their overall satisfaction.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR